| Study Protocol and Statistical Analysis Plan on Palliative Study |
|---|
| Official Study Title: |
| The Effect of Structured Breathing Exercises on Pain, Dyspnea, and Functionality in Terminal |
| Stage Cancer Patients Receiving Palliative Care |
| NCT Number: |
| Pending |
| Document Type: |
| [Study Protocol and Statiscal Analysis] |
| Principal Investigator: |
| Fatma Nur Yildiz Yildirim, PT, MSc |
| Department of Physiotherapy and Rehabilitation |
| Istanbul Atlas University, Turkey |
| nttps://orcid.org/0009-0009-7607-7446 |
| Date of the Document: |
| August 07, 2025 |
| Study Site: |
| Eyupsultan State Hospital, Istanbul, Turkey |
| Study Design: |
| - Interventional, randomized controlled trial (RCT) |
| Two-arm parallel design (Intervention vs. Control) |
| - Single-blinded (evaluator) |
| Study Population: |
| - Total of 39 terminal-stage cancer patients receiving palliative care |

- Intervention group (n = 22), Control group (n = 17)

## Study Protocol and Statistical Analysis Plan on Palliative Study **Inclusion Criteria:** - Age >18 years - Terminal stage cancer diagnosis - Receiving inpatient palliative care - Able to provide consent or have a legal representative **Exclusion Criteria:** - Cognitive impairment preventing exercise compliance - Severe respiratory instability **Intervention Description:** -The intervention group received structured breathing exercises consisting of pursed-lip breathing, diaphragmatic breathing, respiratory control, relaxation breathing exercises, and slow, deep breathing, once a day for 5 days, for an average of 15 minutes. Exercises administered by a physiotherapist. Conducted once daily for 5 consecutive days **Control Group:** - Receives standard palliative care and an informational booklet that describing breathing exercises. **Primary Outcomes:** 1. Pain level (measured by Visual Analog Scale - VAS) 2. Dyspnea (measured by Cancer Dyspnea Scale - CDS) **3.** Functionality (measured by ESAS-r functional subscale)

## **Secondary Outcomes:**

- SpO2, pulse rate, hemoglobin, leukocyte, platelet, CRP levels

## Study Protocol and Statistical Analysis Plan on Palliative Study

